CLINICAL TRIAL: NCT03626285
Title: Institutional Protocol of Bone Marrow Transplantation Using CD34-Selected Peripheral Blood Stem Cells From Related Haploidentical or Unrelated Donors for Treatment of Malignant and Nonmalignant Disorders
Brief Title: Bone Marrow Transplantation Using CD34-Selected Stem Cells From Related or Unrelated Donors in Treating Participants With Cancer or Other Disorders
Status: Available | Type: Expanded Access
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Eneida Nemecek, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: IRB00010804; NCI-2018-00556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2020-02357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00010804 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2018-06-27; First posted 2018-08-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Benign Neoplasm; Bone Marrow Transplantation Recipient; Hematopoietic Cell Transplantation Recipient; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Bone Marrow Transplantation; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Procedure: Bone Marrow Transplantation — Undergo BMT
  Other Names: BMT; Bone Marrow Grafting; Bone marrow transplant; Marrow Transplantation
Device: CliniMACS CD34 Reagent System — CD34 selection ex vivo
Procedure: Peripheral Blood Stem Cell Transplantation — Receive CD34-selected peripheral blood stem cells from related or unrelated donors
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation

SUMMARY:
This expanded access protocol studies bone marrow transplantation using CD34-selected stem cells from related or unrelated donors in treating participants with cancer or other disorders. Stem cells collected from the donor will be processed using a new device called CliniMACS CD34 Reagent System which marks the blood cells collected from the donor with a special protein called "antibody" that tags only the donor stem cells, sorting out other cells of the blood and immune system. This is done to remove, at least partially, some of the T cells. T cells are the cells in the blood that work as scavengers of the immune system deciding what belongs and what does not. These cells can sometimes cause rejection of the donor graft or a condition called graft-versus host disease (GVHD), where the donor cells can attack the body of the recipient. A bone marrow transplantation using CD34-selected stem cells may reduce the risk of these unwanted side effects of transplant as much as possible.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide a source of CD34-selected stem cells for patients with malignant and nonmalignant disorders undergoing bone marrow transplantation from haploidentical (human leukocyte antigen [HLA]-mismatched) related donors or HLA-compatible unrelated donors

SECONDARY OBJECTIVES:

I. Monitoring the safety of the CD34-selected stem cells for the recipient, as measured by adverse events related to stem cell infusion, incidence of engraftment of neutrophils and platelets, incidence of acute and chronic GVHD, and one year overall survival, disease-free survival, and primary disease recurrence.

OUTLINE:

Donor stem cells undergo CD34 selection ex vivo using the CliniMACS CD34 Reagent System using standard operating procedures (SOPs) from the manufacturer. Recipients undergo standard of care preparative regimen, bone marrow transplantation with CD34-selected peripheral blood stem cells via infusion over 1 to 2 hours on day 0, and then receive standard of care GVHD prophylaxis.

After completion of study treatment, recipients are followed up at least once weekly while inpatient until transplant day 100, every 1-3 months for the first year and yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant or nonmalignant diseases that can benefit from alternative stem cell transplantation according to institutional standard practice guidelines
* Patients lacking a healthy human leukocyte antigen (HLA)-identical related donor and having one of the following alternative donor sources:

  * HLA-haploidentical related (HLA antigen genotypic match >= 4/8 and <= 7/8) or
  * Unrelated donor that is HLA matched at >= 7/8 HLA antigen loci
* The selected donor must also be:

  * Able to receive granulocyte colony-stimulating factor (G-CSF, filgrastim) and undergo apheresis either through placement of peripheral or temporary central venous catheter, based on institutional guidelines for peripheral blood stem cell collection
  * Meet all institutional standard criteria for clearance for peripheral stem cell collection
* Recipients must meet institutional treatment standards based on pre-transplant evaluations including:

  * Adequate major organ functions
  * Free of major systemic infections
  * Not pregnant, if female of childbearing age (post-pubertal)
* Recipient (if >= 18 years) or their parent/legal guardian (if < 18 years) must be able to sign the informed consent form for the treatment plan; assent will be obtained from recipients 7-17 years of age, in accordance to our institutional guidelines

Exclusion Criteria:

* Patients not meeting clearance criteria for bone marrow transplantation (BMT) based on standard institutional guidelines
* Presence of anti-HLA antibodies against donor antigens in a recipient or anti-HLA antibodies against recipient antigens in a donor
* Known allergy to murine (mouse) protein or iron-dextran

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Eneida Nemecek, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States